CLINICAL TRIAL: NCT07181317
Title: WAMIF: Prospective Study in Young Women Presenting Acute Myocardial Infarction in France: Clinical, Morphological and Biological Descriptive Analysis: Cohort Follow up
Brief Title: WAMIF: Prospective Study in Young Women Presenting Acute Myocardial Infarction: Cohort Follow up
Acronym: WAMIF-suivi
Status: Recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-04
Record Dates: First submitted 2025-09-08; First posted 2025-09-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction, Acute
MeSH Terms: conditions — Myocardial Infarction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- WAMIF patients: All patients who participated in the WAMIF study (NCT 03073447) and wish to continue follow-up in the present "WAMIF-suivi" study.
  Interventions: Other: Questionnaires; Other: Major events

INTERVENTIONS:
Other: Questionnaires — Assessment of stress and anxiety and quality of life after myocardial infarct:
  * Stress score: Perceived Stress Scale-4 (PSS-4)
  * Anxiety score: Generalized Anxiety Disorder-7 (GAD-7)
  * Depression score: Patient Health Questionnaire-9 (PHQ-9)
  * Quality of life scores: European Quality of Life-5 Dimensions (EQ-5D) and 12-Item Short-Form General Health Survey (SF-12)
Other: Major events — Collection of information related to major events occurring since inclusion in the WAMIF study

SUMMARY:
The WAMIF study was conducted from 2017 to 2019, including 314 patients in 30 French research centers spread across metropolitan France. It systematically collected the clinical, morphological, and biological characteristics of myocardial infarction cases affecting women under 50 years of age and assessed their short-term (in-hospital) and medium-term (12-month) prognosis. Extending the follow-up beyond 12 months for this first study would provide fundamental data for understanding and improving the care of these patients.

DETAILED DESCRIPTION:
The WAMIF study was conducted from 2017 to 2019, including 314 patients in 30 French research centers spread across metropolitan France. It systematically collected the clinical, morphological, and biological characteristics of myocardial infarction cases affecting women under 50 years of age and assessed their short-term (in-hospital) and medium-term (12-month) prognosis. The main results were: a particularly high incidence of modifiable risk factors affecting 86% of patients, with smoking being the primary cause in 75% of them.The clinical presentation found chest pain in more than 90% of cases. The pathophysiological forms of acute coronary syndrome identified the culprit artery in 90% of cases, a form without obstruction (MINOCA) was found in 17.8% of ST segment elevation infarctions (STEMI), spontaneous dissection in 14.6% of STEMI and 16.3% of NSTEMI.At 12 months, follow-up showed no cardiovascular deaths and two deaths related to neoplastic causes. At the end of this follow-up, 90% had no events. Compared to existing studies, these event rates are extremely low. Extending the follow-up beyond 12 months for this first study would provide fundamental data for understanding and improving the care of these patients. The secondary objective is the evaluation of the quality of life and mental health of women who have had an MI before the age of 50 years at a distance from the acute event.

ELIGIBILITY:
All patients who participated in the WAMIF study (research registration number with the French Ministry of Health : 2015-A01263-46 / Protocol registration with Clinical Trials NCT03073447) and wish to continue follow-up in the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 314 women who had a myocardial infarction at less than 50 years, included in the WAMIF study conducted from 2017 to 2019 in 30 French research centers.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | 5 to 10 years after the participation in WAMIF study
  Number of patient who died from any cause since their participation in WAMIF study
Cardiovascular death | 5 to 10 years after the participation in WAMIF study
  Number of patient who died from cardiovascular cause since their participation in WAMIF study
Stent thrombosis | 5 to 10 years after the participation in WAMIF study
  Number of patient who had stent thrombosis since their participation in WAMIF study
Stroke | 5 to 10 years after the participation in WAMIF study
  Number of patient who had stroke since their participation in WAMIF study
Recurrent myocardial infarct | 5 to 10 years after the participation in WAMIF study
  Number of patient who had recurrent myocardial infarct since their participation in WAMIF study
Emergency revascularization | 5 to 10 years after the participation in WAMIF study
  Number of patient who had emergency revascularization since their participation in WAMIF study
Major bleeding | 5 to 10 years after the participation in WAMIF study
  Number of patient who had since major bleeding their participation in WAMIF study
Emergency hospitalization for heart failure | 5 to 10 years after the participation in WAMIF study
  Number of patient who had emergency hospitalization for heart failure since their participation in WAMIF study
Emergency department visit | 5 to 10 years after the participation in WAMIF study
  Number of patient who went to emergency department since their participation in WAMIF study

SECONDARY OUTCOMES:
Stress score | 5 to 10 years after the participation in WAMIF study
  Perceived Stress Scale 4 items. It provides a total score (range 10-50, from worst to best) to assess the state of stress perceived by the patient
Anxiety score | 5 to 10 years after the participation in WAMIF study
  Generalized Anxiety Disorder 7 items. It provides a total score to evaluate patient anxiety (range 0 to 21: 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety)
Depression score | 5 to 10 years after the participation in WAMIF study
  Patient Health Questionnaire 9 items. It provides a total score (range 0-27, 1-4 minimal depression; 5-9 mild depression; 10-14 moderate depression; 15-19 moderately severe depression; 20-27 severe depression) to diagnose and measure severity of depression.
Quality of life score | 5 to 10 years after the participation in WAMIF study
  European Quality of Life 5 Dimensions. It provides a total score (range 0-100, from worst to the best) to evaluate the generic quality of life
Quality of life score | 5 to 10 years after the participation in WAMIF study
  12 Item Short Form General Health Survey. It determines a respondent's profile in eight fields: physical function, physical role, physical pain, general health, vitality, social functioning, emotional role, and mental health

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane MANZO SILBERMAN, MD, Principal Investigator — Hôpital de la Pitié-Salpêtrière, APHP
Locations (1):
- Hôpital de la Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No